CLINICAL TRIAL: NCT02449447
Title: European Comparative Effectiveness Research on Internet-based Depression in Sweden (E-compared) Treatment). A Randomized Controlled Trial Comparing Blended Internet and Face-to-face CBT Against Treatment as Usual
Brief Title: Blended Depression Therapy: Cognitive Behaviour Therapy Face-to-face and Via Internet
Acronym: E-compared
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-compared
Record Dates: First submitted 2015-03-30; First posted 2015-05-20 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorders
Keywords: Major Depressive Disorder (MDD); Blended treatment; Cognitive behavior Therapy (CBT); Face-to-face; internet-based treatment
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blended treatment (Experimental): 10 weeks of four face-to-face Cognitive behavioral therapy sessions and internet-based CBT as a complement and support to the four sessions.
  Interventions: Behavioral: Cognitive behavioral therapy
- Treatment as usual (Active Comparator): Usual course of antidepressants and management in primary care (e.g medication and supportive counselling).
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — CBT based on behavioral activation and cognitive therapy techniques including homework
  Arms: Blended treatment
Other: Treatment as usual — Treatment as usual in primary care including antidepressants and counselling
  Arms: Treatment as usual

SUMMARY:
To asses the clinical effectiveness of blended cognitive behavior therapy (CBT): face-to-face and internet-based treatment for adults with Major Depressive Disorder (MDD) in primary care compared to treatment as usual.

DETAILED DESCRIPTION:
The study is part of a EU-project. Participants are recruited via regular routes from primary care settings. Following the Mini International Neuropsychiatric Interview (M.I.N.I.) participants will be randomly allocated to either blended treatment for 10 sessions/weeks or to treatment as usual. We will include 150 participants in total.

ELIGIBILITY:
Inclusion Criteria:

* depressive symptoms according to DSM-IV
* have access to a computer with internet connection
* have good knowledge of the Swedish language

Exclusion Criteria:

* recent (during last 6 weeks) change in psychiatric medication
* presently in any other psychological treatment
* severe depression
* suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology Self-Report (QIDS | Change from baseline in symptoms of depression. Time Frame: 0, 3, 6 and 12 months
  Symptoms of depression measured by the QIDS. The QIDS is a questionnaire that screens for depressive symptoms and assesses depression severity.

SECONDARY OUTCOMES:
EuroQol-5D (EQ-5D-5L) | Time Frame: 0, 3, 6 and 12 months
  Quality of life will be assessed with the EQ-5D-5L (EuroQol). The EQ-5D-5L is a self-report questionnaire which measures health related quality of life.
Client Satisfaction Questionnaire (CSQ-8) | Time Frame: 3 months (post treatment)
  Patient's satisfaction with the treatment is assessed with Client Satisfaction Questionnaire (CSQ-8)
Credibility and Expectancy Questionnaire (CEQ) | Time Frame: 3 months (post treatment)
  Patients' expectancy of treatment will be assessed with the credibility and expectancy questionnaire (CEQ)
System Usability Scale (SUS) | Time Frame: 3 months (post treatment)
  Satisfaction with the internet platform will be evaluated with the system usability scale (SUS)
Patient Health Questionnaire (PHQ-9) | Time Frame: 0, 3, 6 and 12 months
  The PHQ-9 is a nine-item mood module that can be used to screen and to diagnose patients with depressive disorders.
Working Alliance Inventory (WAI-SF) | Time Frame: 0 months ( three weeks after started treatment)
  The therapeutic alliance between therapists and patient will be assessed with the short version of the Working Alliance Inventory (WAI-SF).
Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TIC-P) | Time Frame: 0, 3, 6 and 12 months
  Health service uptake and production loss due to illness will be measured with the Trimbos and iMTA Questionnaires on Costs Associated with Psychiatric Illness (TiC-P)

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Riper, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Doukani A, Quartagno M, Sera F, Free C, Kakuma R, Riper H, Kleiboer A, Cerga-Pashoja A, van Schaik A, Botella C, Berger T, Chevreul K, Matynia M, Krieger T, Hazo JB, Draisma S, Titzler I, Topooco N, Mathiasen K, Vernmark K, Urech A, Maj A, Andersson G, Berking M, Banos RM, Araya R. Comparison of the Working Alliance in Blended Cognitive Behavioral Therapy and Treatment as Usual for Depression in Europe: Secondary Data Analysis of the E-COMPARED Randomized Controlled Trial. J Med Internet Res. 2024 May 31;26:e47515. doi: 10.2196/47515. PMID 38819882
- [Derived] van Genugten CR, Schuurmans J, Hoogendoorn AW, Araya R, Andersson G, Banos R, Botella C, Cerga Pashoja A, Cieslak R, Ebert DD, Garcia-Palacios A, Hazo JB, Herrero R, Holtzmann J, Kemmeren L, Kleiboer A, Krieger T, Smoktunowicz E, Titzler I, Topooco N, Urech A, Smit JH, Riper H. Examining the Theoretical Framework of Behavioral Activation for Major Depressive Disorder: Smartphone-Based Ecological Momentary Assessment Study. JMIR Ment Health. 2021 Dec 6;8(12):e32007. doi: 10.2196/32007. PMID 34874888
- [Derived] Vernmark K, Hesser H, Topooco N, Berger T, Riper H, Luuk L, Backlund L, Carlbring P, Andersson G. Working alliance as a predictor of change in depression during blended cognitive behaviour therapy. Cogn Behav Ther. 2019 Jul;48(4):285-299. doi: 10.1080/16506073.2018.1533577. Epub 2018 Oct 29. PMID 30372653
- [Derived] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181